CLINICAL TRIAL: NCT02268942
Title: A Prospective, Single-Arm, Multi-Center Study in Collaboration With INTERMACS to Evaluate the Thoracotomy Implant Technique of the HeartWare™ HVAD™ System in Patients With Advanced Heart Failure
Brief Title: HW006 LATERAL Thoracotomy
Acronym: HVAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: INTERMACS (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HW006 Thoracotomy
Record Dates: First submitted 2014-10-16; First posted 2014-10-20 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Left Sided Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Thoracotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- HeartWare HVAD via Thoracotomy (Experimental): HeartWare HVAD implanted via thoracotomy
  Interventions: Device: HeartWare HVAD; Procedure: Thoracotomy

INTERVENTIONS:
Device: HeartWare HVAD — Implant of HeartWare HVAD via thoracotomy implant technique
Procedure: Thoracotomy — Thoracotomy implant technique

SUMMARY:
This is a prospective, multi-center,single-arm study that will evaluate the thoracotomy implant technique in up to 145 subjects implanted via thoracotomy with the HeartWare HVAD System and enrolled in the Interagency Registry for Mechanically Assisted Circulatory Support (Intermacs®) protocol and database.

All participating centers are current INTERMACS® sites in good standing and follow the INTERMACS® protocol and procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥19 years of age at time of informed consent to participate in the Intermacs® registry.
2. Subject receives a HeartWare HVAD (The device should be the subject's first VAD implant).
3. Subject signed an Intermacs® informed consent if required by local IRB policy.
4. Subject signed a HeartWare informed consent.

Exclusion Criteria:

1. Subject is incarcerated (prisoner).
2. Subject did not sign the informed consent at sites where waiver of consent was not granted.
3. Body Surface Area (BSA) < 1.2 m^2.
4. Prior cardiac transplant or cardiomyoplasty.
5. Subject is receiving a BiVAD.
6. Subject is receiving the device as an RVAD.
7. Subject data is generated from non- Intermacs® centers.
8. Pediatric subjects (< 19 years of age).
9. Subjects who receive a temporary LVAD
10. Subjects whose device strategy is listed as "Destination Therapy" at the time of implant.
11. Severe Right Heart failure
12. Aortic insufficiency or mechanical aortic valve.
13. Planned concomitant procedure (e.g.valve repair or replacement, CABG, septal defect repair).
14. Known LV Thrombus.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2014-11; Primary Completion 2016-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (25):
  - The University of Alabama, Birmingham, Alabama
  - Stanford University School of Medicine, Palo Alto, California
  - UC San Diego, San Diego, California
  - UCSF Medical Center, San Francisco, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Tampa Transplant Institute/Tampa General Hospital, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - IU Health Methodist, Indianapolis, Indiana
  - St. Vincent Hospital, Indianapolis, Indiana
  - Jewish Hospital - Rudd Heart and Lung Institute, Louisville, Kentucky
  - John Ochsner Heart & Vascular Institute, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Mayo Rochester - St. Mary's Hospital, Rochester, Minnesota
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
- St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] McGee E Jr, Danter M, Strueber M, Mahr C, Mokadam NA, Wieselthaler G, Klein L, Lee S, Boeve T, Maltais S, Pretorius GV, Adler E, Vassiliades T, Cheung A. Evaluation of a lateral thoracotomy implant approach for a centrifugal-flow left ventricular assist device: The LATERAL clinical trial. J Heart Lung Transplant. 2019 Apr;38(4):344-351. doi: 10.1016/j.healun.2019.02.002. PMID 30945636
- [Derived] Wieselthaler GM, Klein L, Cheung AW, Danter MR, Strueber M, Mahr C, Mokadam NA, Maltais S, McGee EC Jr. Two-Year Follow Up of the LATERAL Clinical Trial: A Focus on Adverse Events. Circ Heart Fail. 2021 Apr;14(4):e006912. doi: 10.1161/CIRCHEARTFAILURE.120.006912. Epub 2021 Apr 19. PMID 33866829
- [Derived] Mahr C, McGee E Jr, Cheung A, Mokadam NA, Strueber M, Slaughter MS, Danter MR, Levy WC, Cheng RK, Beckman JA, May DM, Ismyrloglou E, Tsintzos SI, Silvestry SC. Cost-Effectiveness of Thoracotomy Approach for the Implantation of a Centrifugal Left Ventricular Assist Device. ASAIO J. 2020 Aug;66(8):855-861. doi: 10.1097/MAT.0000000000001209. PMID 32740343

RESULTS

PARTICIPANT FLOW:
Groups:
- Per Protocol Population: Subjects meeting eligibility criteria and received an HVAD implanted via thoracotomy.
Period: Overall Study
Arm/Group | Per Protocol Population
Started | 144
Completed | 144
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Per Protocol Population
Number analyzed (Participants) | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 subject refused to answer
  Participants
    number analyzed (Participants) | 143
    Female | 32
    Male | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 132
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 30
  White | 90
  More than one race | 3
  Unknown or Not Reported | 11
Region of Enrollment [Number; unit: participants]
  Canada | 3
  United States | 141
Height [Mean (Standard Deviation); unit: centimeters] | 175.2 (8.8)
Weight [Mean (Standard Deviation); unit: kilograms] | 83.5 (18.8)
Body Mass Index [Mean (Standard Deviation); unit: kilograms per meters squared] | 27.1 (5.1)
Body Surface Area [Mean (Standard Deviation); unit: meters squared] | 2.0 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Subject is Alive on Original Device, Transplanted, or Explanted for Recovery at 6 Months
Description: * Alive on the originally implanted device at six months, and the subject has not had a stroke with a modified Rankin Scale ≥ 4 (assessed ≥ three months post-stroke event); or
  * Transplanted by Month 6, and the subject has not had a stroke with a modified Rankin Scale
    ≥ 4 (assessed ≥ three months post-stroke event); or
  * Explanted for recovery by Month 6, and the subject has not had a stroke with a modified Rankin Scale ≥ 4 (assessed ≥ three months post-stroke event).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Per Protocol Population
Number analyzed (Participants) | 143
Participants | 128
Statistical Analysis 1: Comparison: Per Protocol Population; Success at six months is estimated to be 86% compared to a performance goal of 77.5%. Using an exact binomial test, with a one-sided alpha of 0.05, and 80% Power, a sample size of 145 implanted subjects was planned. Success will be met if the lower bound of the upper one-sided exact 95% confidence interval is greater than 77.5%; Test type: Other; p = 0.0003, Exact Binomial

2. Secondary Outcome: Mean Length of Initial Hospital Stay
Description: Mean length of initial hospital stay including both acute care (ICU/CCU) and step-down Care time
Time Frame: Initial Hospital Stay
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Per Protocol Population
Number analyzed (Participants) | 144
days | 17.8 (11.7)
Statistical Analysis 1: Comparison: Per Protocol Population; The secondary endpoint is an improvement in the mean length of initial hospital stay (initial recovery and step down unit), which is calculated by considering the number of days in acute care (ICU/CCU) plus the number of days in intermediate/step-down care, comprising the total number of days post-implant to discharge. This secondary endpoint will be calculated using an upper tail one-sided t-test at 0.05 level of significance compared to 26.1 days for median sternotomy patients; Test type: Other; p < 0.0001, t-test, 1 sided

ADVERSE EVENTS:
Description: Intermacs Categories used for collection.
Arm/Group | Per Protocol Population
All-Cause Mortality (participants affected / at risk) | 20/144
Serious Adverse Events (participants affected / at risk) | 134/144
Other Adverse Events (participants affected / at risk) | 44/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Per Protocol Population (N=144)
Major Bleeding (Blood and lymphatic system disorders) | 46 (96)
Cardiac Arrhythmia (Cardiac disorders) | 57 (85)
Device Malfunction/Failure and/or Pump Thrombus (Product Issues) | 42 (83)
Hemolysis (Blood and lymphatic system disorders) | 60
Infection (Infections and infestations) | 66 (130)
Myocardial Infarction (Cardiac disorders) | 0 (0)
Neurological Dysfunction (Vascular disorders) | 38 (56)
Right Heart Failure (Cardiac disorders) | 53
Hepatic Dysfunction (Hepatobiliary disorders) | 3 (3)
Hypertension (General disorders) | 10
Pericardial Fluid Collection (General disorders) | 5 (5)
Psychiatric Episode (Psychiatric disorders) | 8 (8)
Renal Dysfunction (Renal and urinary disorders) | 18 (20)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 18 (23)
Arterial Non-CNS Thromboembolism (Cardiac disorders) | 0 (0)
Venous Thromboembolism (Cardiac disorders) | 6 (6)
Wound Dehiscence (General disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Per Protocol Population (N=144)
Other (General disorders) | 44 (99) — "Other" is an adverse event term category in the Intermacs registry and no additional data was provided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, the contract allows the principal investigator to publish their data after the release of the multi-center publication (or one year after the conclusion of the study if no multi-center publication is submitted) following the sponsor review for (a) disclosure of confidential information, and (b) information that would impair the sponsor's ability to obtain patent protection.

DOCUMENTS (2):
  • Study Protocol (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT02268942/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT02268942/SAP_001.pdf